CLINICAL TRIAL: NCT05604352
Title: Extended Phase 2 Product Evaluation Single Sample Study - To Evaluate the Safety of the DiaSole Insole for Use on Patients With Diabetic Foot Ulcers
Brief Title: Safety Evaluation of the DiaSole Insole With Diabetic Foot Ulcers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaydiar Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVT001_Protocol
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single sample, no randomisation, no blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main study (Experimental): Study to investigate the safety and clinical efficacy of the DiaSole insole.
  Interventions: Device: DiaSole

INTERVENTIONS:
Device: DiaSole — Diabetic ulcer offloading insole

SUMMARY:
Offloading plays an important part Diabetic foot ulcers healing. The modular design of the DiaSole would allow the offloading cavity to be changed in line with the changing ulcer dimensions. It may be possible to use the DiaSole for other causes of neuropathic foot ulcerations (such as rheumatoid arthritis), but the safety of the insole needs assessing first. There is already evidence to support the use of offloading insoles in the healing and prevention of pressure ulcers, DiaSole may be an improved insole for this purpose.

DETAILED DESCRIPTION:
DiaSole is an insole developed to aid the treatment of diabetic foot ulcers through offloading. Offloading (reducing pressure) plays an integral role in the treatment of diabetic ulcers. DiaSole is modular in construction comprising of many 'cells', which can be individually removed to create the offloading cavity.

This study aims to evaluate the safety of DiaSole with diabetic patients who have superficial ulcers. The ulcer severity of patients included will not involve tendon, capsule or bone, or will be pre or post ulceration and have healed skin integrity (Texas wound classification 1A and 0A respectively).

The study will be conducted within Hywel Dda University Health Board (HDUHB) Podiatry services. Participants will be seen in clinic by the podiatrists emplyed within HDUHB. The patients who consent to take part will be issued a DiaSole insole as part of their usual care and under guidance of the podiatrist. The participants will be instructed to use the DiaSole as part of their ulcer offloading, for an 8-week period.

The primary outcome of this study is to assess the safety of the DiaSole insole with patients who have diabetic neuropathy and are at risk of a pressure ulcer in the feet and/or who have a superficial pressure ulcer. All adverse events and serious adverse events will be documented and used to assess the safety of DiaSole.

During the 8-week period the participants will have photographs taken of their pressure ulcer sites so that any changes to its size can be monitored. The depth of the ulcer will also be measured using a probe. The ulcer dimensions will be monitored as a secondary outcome and data will be collected during the first appointment, then again at weeks 1,2,3,4 and then week 8.

An evaluation form will also be used to capture clinician and patient feedback regarding acceptability at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Capacity to consent
* UK Shoe size 3-11
* Diagnosis of Diabetes
* Sensory neuropathy (lack of perception of 10g monofilament in one or more sites of the feet)
* Active foot ulceration (plantar aspect), grade 1a using the University of Texas wound grading system (grade 1a)
* Appropriate footwear (which has room to safely accommodate the DiaSole insole)
* At risk of ulceration or re-ulceration (Grade 0A)

Exclusion Criteria:

* Patients who are non-concordant and do not have appropriate footwear that could house the DiaSole insole
* Clinical signs of or confirmed active infection (soft tissue or osteomyelitis)
* History of or active Charcot foot or severe foot deformity
* Amputation
* Critical limb ischemia or diagnosed moderate to severe peripheral arterial disease
* Inappropriate footwear (does not accommodate the DiaSole insole)
* Visual impairment (cannot see feet and footwear properly)
* Sensory neuropathy of the upper limbs/hands
* History of drug and alcohol abuse• Have known contraindications to the materials used in the product insoles. Allergies to cotton or silicone
* Have an infectious disease, which may pose as a potential risk to the researchers and clinicians
* Are enrolled into another study
* Unable to attend regular hospital visits - e.g. housebound
* Are unwilling to take part in the study
* Are currently enrolled in any other research
* Individuals who do not adequately understand verbal explanations of written information in English, unless there is access to a qualified translator
* Are not suitable for the evaluation, according to the podiatrist's or nurse's clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-04-28 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the safety of the DiaSole insole | 8-weeks per patient
  Recording adverse events

SECONDARY OUTCOMES:
Clinical efficacy of DiaSole insole | 8-weeks per patient
  Assessing wound closure area (mm2)
acceptability of DiaSole to health care professionals (HCPs) | 8-weeks per patient
  Survey based feedback from HCPs

IPD SHARING:
Plan to Share IPD: No
No patient identifiable information will be shared outside of the direct care team or the research team.